CLINICAL TRIAL: NCT00992238
Title: A Relative Bioavailability Study of 100 mg Flavoxate Hydrochloride Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R03155
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Flavoxate

ARMS (2):
- Flavoxate Hydrochloride Tablets, 100mg (Experimental)
  Interventions: Drug: Flavoxate Hydrochloride Tablets, 100mg
- Urispas® Tablets, 100mg (Active Comparator)
  Interventions: Drug: Urispas® Tablets, 100mg

INTERVENTIONS:
Drug: Flavoxate Hydrochloride Tablets, 100mg
  Arms: Flavoxate Hydrochloride Tablets, 100mg
Drug: Urispas® Tablets, 100mg
  Arms: Urispas® Tablets, 100mg

SUMMARY:
The purpose of this study is to compare the relative bioavailability of Flavoxate Hydrochloride tablets 100mg manufactured by Paddock Laboratories, Inc., with that of Urispas® tablets 100mg by SmithKline Beecham Pharmaceuticals under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by lack of clinically significant abnormalities in health assessment performed at screening

Exclusion Criteria:

* Positive test results for HIV or Hepatitis B or C
* History of allergy or sensitivity to Flavoxate hydrochloride or related drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd, Fargo, North Dakota, United States